CLINICAL TRIAL: NCT01900743
Title: Activity and Safety of Regorafenib in Patients With Metastatic Soft Tissue Sarcoma Previously Treated With Anthracycline-based Chemotherapy : a Multinational, Randomized, Phase II, Placebo-controlled Trial
Brief Title: Phase II Study of Regorafenib in Metastatic Soft Tissue Sarcoma
Acronym: REGO-SARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REGO-SARC-1214; 2012-005743-24 (EudraCT Number)
Record Dates: First submitted 2013-07-09; First posted 2013-07-16 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Sarcoma
Keywords: Sarcoma; Metastatic; Regorafenib
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Regorafenib (160 mg/d) once daily for 3 weeks on / 1 week off plus Best Supportive Care (BSC) until progression (according to RECIST 1.1), intolerance or consent withdrawal.
  Interventions: Drug: Regorafenib
- Arm B (Placebo Comparator): Placebo plus BSC until progression (according to RECIST 1.1) or unacceptable toxicity. Patients who have received placebo may be offered open-label regorafenib (cross-over option) after objective tumor progression
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib — Regorafenib (160 mg/d) once daily for three weeks on / one week off plus Best Supportive Care (BSC)until progression (according to RECIST 1.1), intolerance or consent withdrawal.
  Other Names: stivarga
  Arms: Arm A
Drug: Placebo — Placebo plus BSC until progression (according to RECIST 1.1) or unacceptable toxicity. Patients who have received placebo may be offered open-label regorafenib (cross-over option) after objective tumor progression
  Arms: Arm B

SUMMARY:
This is an international (France, Austria and Germany), randomized, double-blind, placebo-controlled, phase II study to evaluate the efficacy and safety of regorafenib in patients with histologically proven metastatic and/or unresectable Soft Tissue Sarcoma (STS) after failure or intolerance to doxorubicin (or other anthracycline).

Five cohorts will be defined:

Cohort A: Liposarcoma Cohort B: Leiomyosarcoma Cohort C: Synovial sarcoma Cohort D: other sarcomas (see Appendix C) Cohort E: Leiomyosarcoma, Synovial sarcoma and other sarcomas listed in Appendix C previously treated with pazopanib Approximately 226 patients who meet the eligibility criteria will be randomly assigned in a 1:1 ratio to one of the treatment groups.

DETAILED DESCRIPTION:
The standard of care for metastatic soft tissue sarcoma is doxorubicin +/- ifosfamide. After failure or intolerance to doxorubicin, there is no standard of care. In Europe, two are currently approved for the treatment of soft tissue sarcoma after failure/intolerance to doxorubicin: trabectedin (Yondelis®) for all histological subtype and pazopanib (Votrient ®) for all subtypes excluding liposarcomas. Nevertheless, none of these drugs improve the overall survival over placebo.

The study is composed of 3 periods:

1. A Screening Period,
2. A Treatment Period,
3. And a Survival Follow-up Period. Patients randomized to be treated with regorafenib will receive the treatment orally for 3 weeks of every 4 week (28 days) cycle (ie, 3 weeks on/1 week off).

Patients randomized to the placebo arm will be treated for 3 weeks of every 4 weeks cycle (ie, 3 weeks on/1 week off).

In addition to the regorafenib and placebo treatments, patients will receive best supportive care. Best supportive care includes any method to preserve the comfort and dignity of the patients and excludes any disease-specific anti-neoplastic therapy such as any kinase inhibitor,chemotherapy, radiation therapy, or surgical intervention.

Patients receiving placebo, who experience disease progression may be offered open-label regorafenib(cross-over option).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histological documentation of soft tissue sarcoma (including uterus)with available Formalin Fixed Paraffin Embedded (FFPE) blocks. Eligible soft tissue sarcomas are non-adipocytic soft tissue sarcomas
* Prior treatment with doxorubicin or other anthracycline. Moreover, patients eligible in the Cohort E must have received pazopanib
* Metastatic disease not amenable to surgical resection with curative intent
* Documentation of progression within the last 6 months
* Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST 1.1.
* Performance status ≤1(ECOG)
* Life expectancy ≤ 3 months
* Adequate bone marrow, renal, and hepatic function:
* INR/PTT ≤1.5 x ULN Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring will be performed until INR/PTT is stable.
* Women of childbearing potential and male patients must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy.
* Recovery to NCI-CTCAE v4.0 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure related toxicity (except alopecia, anemia, and hypothyroidism).
* In the assessment of the investigator, patient is able to comply with study requirements
* Signed, IRB-approved written informed consent

Exclusion Criteria:

* More than 3 lines of systemic treatment for metastatic sarcoma
* Histological subtypes listed in Appendix C (especially GIST, osseous sarcoma, embryonal or alveolar rhabdomyosarcoma). Patients with liposarcoma are not eligible in the cohort E
* Primary bone sarcoma
* Prior treatment with regorafenib
* Known history of or concomitant malignancy likely to affect life expectancy in the judgment of the investigator
* Pregnant or breastfeeding patients. Women of childbearing potential must have a pregnancy test performed before start of treatment
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of treatment
* Active cardiac disease including any of the following: Congestive heart failure (NYHA) ≥Class 2, Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension (SBP >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism (within the last 6 months)
* Ongoing infection >Grade 2 according to NCI-CTCAE v4.0
* Known history of human immunodeficiency virus (HIV) infection
* Known history of chronic hepatitis B or C
* Patients with seizure disorder requiring medication
* History of organ allograft
* Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event > Grade 3 within 4 weeks of start of treatment
* Non-healing wound, ulcer, or bone fracture
* Renal failure requiring hemo- or peritoneal dialysis
* Dehydration according to NCI-CTC v 4.0 Grade >1
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation, including lactose
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Inability to swallow, malabsorption condition
* Pleural effusion or ascites that causes respiratory compromise (Grade 2 dyspnea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-06-05 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-Free Survival will be measured from the date of randomization until the date of radiological progression or death (if death occurs before progression).
  Progression-free rate at 3 and 6 months (PFR-3 and PFR-6), time to progression, response rate and duration of response, overall survival according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Growth modulation index | Up to 2 years
  Growth modulation index in patients receiving regorafenib after randomization
Toxicity according to NCI-CTC AE V4.0. | Baseline, every 4 weeks, up to the end of study
  The monitoring of the toxicity of the regorafenib which can have a liver toxicity for exemple.
Progression-free rate at 3 and 6 months (PFR-3 and PFR-6) | At month 3 and at month 6
  According to the RECIST 1.1
Time to progression | Up to 2 years
  According to the RECIST 1.1 Every 4 weeks, Up to 2 years
Overall survival | Up to 2 years
  Time from the date of randomization to the date of death from any cause
Response rate | Up to 2 years
  the proportion of patients with the best overall tumor response of partial response (PR) or complete response (CR) according to RECIST 1.1 guidelines that is achieved during treatment or within 30 days after termination of study medication.
Duration of response | Up to 2 years
  the number of days from the date of first documented objective response of PR or CR, whichever is noted earlier, to first disease progression or death before progression. Patients without progression or death before progression at the time of analysis will be censored at the date of their last tumor assessment.

OTHER OUTCOMES:
Potential predictive factors for regorafenib response. | Up to 2 years
  The monitoring of the factors which can induce a regorafenib response (Formalin fixed, paraffin embedded (FFPE) or fresh frozen tissue samples collected either from the primary tumor or from metastatic sites, or both will be analyzed)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, PhD, Study Director — Centre Oscar Lambret - France; Thomas BRODOWICZ, PhD, Principal Investigator — AKH-Wien - Austria
Locations (25):
- Austria (5):
  - Medizinische Universität Graz, Graz
  - Universitätsklinik für Innere Medizin I, Innsbruck
  - LKH, Klagenfurt
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - AKH-Wien, Vienna
- France (20):
  - Hôpital St Jacques, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre GF Leclercq, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de La Timone, Marseille
  - Centre René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth (ICL), Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penel N, Mir O, Wallet J, Ray-Coquard I, Le Cesne A, Italiano A, Salas S, Delcambre C, Bompas E, Bertucci F, Saada-Bouzid E, Chaigneau L, Chevreau C, Brodowicz T, Decoupigny E, Vanseymortier M, Laroche L, Taieb S, Le Deley MC, Blay JY. A double-blind placebo-controlled randomized phase II trial assessing the activity and safety of regorafenib in non-adipocytic sarcoma patients previously treated with both chemotherapy and pazopanib. Eur J Cancer. 2020 Feb;126:45-55. doi: 10.1016/j.ejca.2019.12.001. Epub 2020 Jan 6. PMID 31918233
- [Derived] Longue M, Cabarrou B, Wallet J, Brodowicz T, Roche H, Boher JM, Delord JP, Penel N, Filleron T. The importance of jointly analyzing treatment administration and toxicity associated with targeted therapies: a case study of regorafenib in soft tissue sarcoma patients. Ann Oncol. 2018 Jul 1;29(7):1588-1593. doi: 10.1093/annonc/mdy168. PMID 29722789
- [Derived] Berry V, Basson L, Bogart E, Mir O, Blay JY, Italiano A, Bertucci F, Chevreau C, Clisant-Delaine S, Liegl-Antzager B, Tresch-Bruneel E, Wallet J, Taieb S, Decoupigny E, Le Cesne A, Brodowicz T, Penel N. REGOSARC: Regorafenib versus placebo in doxorubicin-refractory soft-tissue sarcoma-A quality-adjusted time without symptoms of progression or toxicity analysis. Cancer. 2017 Jun 15;123(12):2294-2302. doi: 10.1002/cncr.30661. Epub 2017 Mar 10. PMID 28295221
- [Derived] Mir O, Brodowicz T, Italiano A, Wallet J, Blay JY, Bertucci F, Chevreau C, Piperno-Neumann S, Bompas E, Salas S, Perrin C, Delcambre C, Liegl-Atzwanger B, Toulmonde M, Dumont S, Ray-Coquard I, Clisant S, Taieb S, Guillemet C, Rios M, Collard O, Bozec L, Cupissol D, Saada-Bouzid E, Lemaignan C, Eisterer W, Isambert N, Chaigneau L, Cesne AL, Penel N. Safety and efficacy of regorafenib in patients with advanced soft tissue sarcoma (REGOSARC): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2016 Dec;17(12):1732-1742. doi: 10.1016/S1470-2045(16)30507-1. Epub 2016 Oct 14. PMID 27751846
- [Derived] Brodowicz T, Liegl-Atzwager B, Tresch E, Taieb S, Kramar A, Gruenwald V, Vanseymortier M, Clisant S, Blay JY, Le Cesne A, Penel N. Study protocol of REGOSARC trial: activity and safety of regorafenib in advanced soft tissue sarcoma: a multinational, randomized, placebo-controlled, phase II trial. BMC Cancer. 2015 Mar 14;15:127. doi: 10.1186/s12885-015-1143-y. PMID 25884155